CLINICAL TRIAL: NCT06170970
Title: Solriamfetol for the Treatment of Fatigue in Patients With Multiple Sclerosis and Excessive Daytime Sleepiness
Brief Title: Solriamfetol for the Treatment of Multiple Sclerosis Fatigue
Acronym: SOLARIMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Multiple Sclerosis Society (Other); Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00295382
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis Fatigue
Keywords: multiple sclerosis; fatigue; daytime sleepiness
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Disorders of Excessive Somnolence | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- solriamfetol then placebo first (Experimental): Four weeks of treatment with solriamfetol followed by one week of washout and four weeks of treatment with placebo
  Interventions: Drug: Solriamfetol; Drug: Placebo
- placebo then solriamfetol first (Experimental): Four weeks of treatment with placebo followed by one week of washout and four weeks of treatment with solriamfetol
  Interventions: Drug: Solriamfetol; Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol — solriamfetol 75 mg daily for 3 days and will increase the dose to 150 mg daily starting on day 4 of the treatment period (total of four weeks)
  Other Names: Sunosi
Drug: Placebo — Four weeks of oral placebo

SUMMARY:
Fatigue is a prevalent and disabling symptom in Multiple Sclerosis (MS), affecting up to 90% of patients. Current treatments, including off-label prescriptions of wake-promoting agents, have shown limited effectiveness. Previous research indicates that these agents may be beneficial specifically for MS patients with concomitant excessive daytime sleepiness. This study uses a randomized, double-blind, placebo-controlled crossover design. Participants will undergo a 10-day lead-in with he medication/placebo, followed by two four-week treatment periods separated by a one-week washout. Outcomes will be measured primarily using the Modified Fatigue Impact Scale (MFIS), with additional exploratory measures collected via a smartphone app that assesses fatigue through keystroke dynamics. This novel approach to fatigue measurement aims to capture real-time variations and provide more granular data than traditional self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 60 years of age, inclusive.
* Medically stable on the basis of physical examination, medical history, and vital signs
* Must meet McDonald 2017 diagnostic criteria for multiple sclerosis based on the PI review of the medical records
* Must complain from fatigue as one of their main symptoms and have a screening MFIS score of 33 or more
* A screening ESS score of 10 or more
* Must be ambulatory (able to walk at least 20 feet using bilateral assistance)
* Must have internet and email access and the ability to use a computer or tablet, or smartphone
* Own an android smartphone or an iphone
* Consent to use a medically acceptable method of contraception for the duration of the study
* Willing and able to comply with the study design schedule and other requirements
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of coronary artery disease or congestive heart failure
* Uncontrolled hypertension at Screening (history of high blood pressure and screening systolic blood pressure >160 or diastolic blood pressure>100)
* A known history of uncontrolled diabetes (the last known hemoglobin A1c level above 7.0%), high BMI (>35), or hyperlipidemia (last known total cholesterol >240 mg/dl, or LDL cholesterol level >160 mg/dl)
* Receiving drugs/treatments that increase blood pressure or heart rate (based on the PI review of the medications/treatments)
* A history of cerebrovascular disease or stroke
* A medical or neurological disorder other than MS, that was associated with excessive sleepiness.
* A history of phenylketonuria or hypersensitivity to the phenylalanine-derived product
* A history of alcohol or drug abuse within the past two years
* A history of psychosis, or bipolar disorder
* A history of cardiac arrythmias
* The use of any product with stimulating or sedating properties, unless they have been on a steady dose for at least a month prior to the screening visit and agree to stay on the same dose over the course of the study
* Use within 14 days of a monoamine oxidase (MAO) inhibitor drug
* Pregnant or lactating
* Use of medications used for the treatment of fatigue (including amantadine, modafinil, armodafinil, and amphetamine-like stimulants) in the past two weeks of the screening visit
* A known history of moderate or severe kidney dysfunction (estimated Glomerular filtration rate of less than 60 mL/min)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) Score | Up to 4 weeks
  MFIS score measured during the last three days of each 4-week medication period. The total score of the MFIS ranges from 0 to 84. Higher scores denote more severe fatigue.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) Score | Up to 4 weeks
  FSS score measured during the last three days of each 4-week medication period. The total score of the FSS ranges from 1 to 7. Higher scores denote more severe fatigue.
Epworth Sleepiness Scale (ESS) Score | Up to 4 weeks
  ESS score measured during the last three days of each 4-week medication period. The total score of the ESS ranges from 0 to 24. Higher scores denote more severe daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators have set a timeline for data availability, commencing one year after the publication of the trial's main findings and extending for a period of five years. This timeframe ensures data relevance while providing ample opportunity for research exploration.
  Access to the data will be governed by a stringent but fair set of criteria. Interested researchers must submit a methodologically sound proposal, which will be evaluated by an independent review panel. This process ensures that the data are used to pursue scientifically valuable and ethically sound objectives.
  Researchers accessing the data must agree to terms that uphold privacy, ensure data security, and prohibit the further sharing of data with third parties.
Supporting Information: Study Protocol, SAP
Time Frame: one year after the publication of the main trial results to 5 years after the publication.
Access Criteria: Researchers accessing the data must agree to terms that uphold privacy, ensure data security, and prohibit the further sharing of data with third parties.